CLINICAL TRIAL: NCT03366545
Title: Observation of Clinical Routine Care for Heart Failure Patients Implanted With BIOTRONIK CRT Devices
Acronym: BIO|STREAM HF
Status: Active, not recruiting | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR021
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
Keywords: cardiac resynchronization therapy; CRT; clinical routine
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy (CRT) — Observation and documentation of routine care for CRT patients

SUMMARY:
The registry is primarily designed to assess outcome, efficacy and residual safety aspects of CRT based on long-term data from an unselected, real-life clinical set-up. Moreover, the observation of the patient status should help to find possible predictors for HF events and to identify areas of improvement for CRT and for CRT device settings.

ELIGIBILITY:
Inclusion Criteria:

* Planned de novo implantation of or upgrade to a CRT system for treatment according to the intended use
* Patient is able to understand the nature of the registry and has provided written informed consent
* Patient is willing and able to use the CardioMessenger and accepts the Home Monitoring concept
* Remote monitoring using the Home Monitoring® platform is planned for the patient

Exclusion Criteria:

* Standard contraindication for CRT
* Already or previously implanted with CRT system
* • Age < 18 years
* Participation in another interventional clinical investigation other than the registry-based trials of BIO|STREAM.HF
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representative population of CRTpatients at clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 3030 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of cardiovascular adverse events | throughout study duration, average of 3.5 years; annual evaluations
  Number of unplanned hospitalization for cardiovascular cause
Number of patient deaths | throughout study duration, average of 3.5 years; annual evaluations
  Number of all-cause mortality
Number of all cause hospitalization | throughout study duration, average of 3.5 years; annual evaluations
  Number of all cause hospitalization
Number of patients with worsening of heart failure events | throughout study duration, average of 3.5 years; annual evaluations
  Number of unplanned hospitalization for worsening of heart failure
Number of patients with cerebrovascular events | throughout study duration, average of 3.5 years; annual evaluations
  Number of cerebrovascular events requiring hospitalization
Number of all adverse device effects | throughout study duration, average of 3.5 years; annual evaluations
  Number of all adverse device effects
Number of all device deficiencies | throughout study duration, average of 3.5 years; annual evaluations
  Number of all device deficiencies
Assessment of patients benefit from CRT | throughout study duration, average of 3.5 years; annual evaluations
  Documentation of NYHA classification [I-IV]
Number of patient deaths with cardiovascular cause | throughout study duration, average of 3.5 years; annual evaluations
  Number of patient deaths with cardiovascular cause
Documentation of LVEF | throughout study duration, average of 3.5 years; annual evaluations
  Left ventricular ejection fraction [%]
Documentation of LVESV | throughout study duration, average of 3.5 years; annual evaluations
  Left ventricular end-systolic volume [ml]

CONTACTS AND LOCATIONS:
Locations (114):
- Australia (7):
  - Canberra Heart Rhythm Foundation, Canberra
  - The Canberra Hospital, Canberra
  - Lyell McEwin Hospital, Elizabeth Vale
  - Liverpool Hospital, Liverpool
  - Sydney Adventist Hospital, Sydney
  - Westmead Hospital, Westmead
  - Westmead Private Hosptial, Westmead
- Austria (3):
  - Kepler Universitätsklinikum, Linz
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - Imelda Ziekenhuis, Bonheiden
  - UZ Brussel, Brussels
  - CHR de la Citadelle - Liège, Liège
- Czechia (3):
  - Nemocnice České Budějovice, České Budějovice
  - Fakultní nemocnice Olomouc, Olomouc
  - Institute for Clinical and Experimental Medicine (IKEM), Prague
- France (23):
  - CHU de Brest, Brest
  - Le Centre Hospitalier Universitaire de CAEN, Caen
  - Centre Hospitalier Louis Pasteur, Chartres
  - CH Saint Philibert, Lomme
  - Centre Hospitalier Lorient, Lorient
  - Hôpital privé Clairval, Marseille
  - Hopital de la Timone (CHU La Timone), Marseille
  - Hôpital Privé / Institute Jaques Cartier, Massy
  - Clinique les Fontaines, Melun
  - CHU Montpellier, Montpellier
  - Clinique du Millenaire, Montpellier
  - Hôpital privé du Confluent, Nantes
  - Hopital Pitie-Salpetriere, Paris
  - Hôpital Haut Lévêque, Pessac
  - Centre Hospitalier de Périgeux, Périgueux
  - Centre Hospitalier Universitaire de Saint-Étienne, Saint-Etienne
  - Centre Hospitalier Mémorial de Saint-Lô, Saint-Lô
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre Hospitalier de Rangueil, Toulouse
  - Clinique Pasteur Toulouse, Toulouse
  - Chru de Tours, Tours
  - CH de Valence, Valence
  - Centre Hospitalier Bretagne Atlantique Prosper Chubert, Vannes
- Germany (19):
  - Städtisches Klinikum St.Georg, Leipzig, Saxony
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - HDZ Bad Oeynhausen, Bad Oeynhausen
  - Maria Heimsuchung - Carita-Klinik Pankow, Berlin
  - Städtisches Klinikum Brandenburg GmbH, Brandenburg
  - Krankenhaus Buchholz und Winsen AöR, Buchholz
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Giessen und Marburg, Giessen
  - KMG Klinikum Güstrow, Güstrow
  - Klinikum der Universität Jena, Jena
  - Bonifatius Hospital Lingen gGmbH, Lingen
  - Universitätsklinikum Schleswig-Holstein (UKSH) - Campus Lübeck, Lübeck
  - Carl-von-Basedow-Klinikum Saalekreis GmbH, Merseburg
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der LMU / Campus Großhadern, München
  - Universitätsklinikum Münster, Münster
  - Städtische Kliniken Neuss -Lukaskrankenhaus- GmbH, Neuss
  - Schüchtermann Klinik, Herzzentrum Osnabrück-Bad Rothenfelde, Rothenfelde
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (4):
  - State Hospital of Cardiology, Balatonfüred
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Semmelweis Medical University, Budapest
  - The University of Pécs, Pécs
- Israel (9):
  - Assuta Medical Center, Ashdod
  - Ben-Gurion University of the Negev, Beersheba
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Chaim Sheba Medical Center, Tel Litwinsky
  - Shamir Medical Center, Ẕerifin
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Policlinico Casilino, Roma
- Japan (7):
  - Kokura Memorial Hospital, Fukuoka
  - Hiroshima Prefectural Hospital, Hiroshima
  - Tokai University Hospital, Kanagawa
  - Kitasato University Hospital, Sagamihara
  - Saitama Medical University International Medical Center, Saitama
  - Juntendo University Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Poland (3):
  - Medical University of Lodz, Lodz
  - Szpital Kliniczny Przemienienia Pańskiego, Poznan
  - The National Cardiology Institute of Stefan Cardinal Wyszynski - National Research Institute, Warsaw
- Portugal (4):
  - Hospital de Santa Cruz, Carnaxide
  - Hospital Espirito Santo de Evora, Evora
  - Hospital de Santa Maria, Lisbon
  - Hospital de Santo António, Porto
- Changi General Hospital, Singapore, Singapore
- Slovakia (3):
  - SÚSCCH, Banská Bystrica
  - NÚSCH Bratislava a.s., Bratislava
  - East-Slovak Cardiology Institute (VUSCH), Košice
- South Africa (6):
  - Mediclinic Panorama Hospital, Cape Town
  - Mediclinic Pietermaritzburg, Pietermaritzburg
  - Mediclinic Midstream, Pretoria
  - Unitas Hospital, Pretoria
  - Gateway Private Hospital, Umhlanga
  - Life Westville, Westville
- Spain (10):
  - Hospital General Universitario de Alicante, Alicante
  - Centro Médico Teknon, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario La Fé, Valencia
  - Hospital Álvaro Cunqueiro, Vigo
- Universitätsspital Zürich, Zurich, Switzerland
- Taiwan (2):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
- United Kingdom (3):
  - St. Peter's Hospital, Chertsey
  - Russells Hall Hospital, Dudley
  - Kettering General Hospital, Kettering

IPD SHARING:
Plan to Share IPD: No
No individual participant data in planned to be shared with other researchers